CLINICAL TRIAL: NCT03908723
Title: Treatment of Macular Edema Caused by Leber's Miliary Aneurysms Using Intravitreal Aflibercept and Peripheral Laser Photocoagulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed M. Abdel Hadi, Assistant Professor ophthalmology Faculty of Medicine, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21526
Record Dates: First submitted 2019-04-07; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Macular Edema Caused by Leber's Miliary Aneurysms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all patients in the study (Experimental)
  Interventions: Other: Panretinal photocoagulation

INTERVENTIONS:
Other: Panretinal photocoagulation — Intravitreal Aflibercept with PRP to the peripheral vascular lesions

SUMMARY:
This study evaluates the effectiveness of intravitreal Aflibercept (IVA) injection therapy, combined with peripheral laser photocoagulation, in the treatment of macular edema caused by Leber's miliary aneurysm. We believe that our study makes a significant contribution to the literature because to our knowledge, it is the first to report cases, in which IVA injection therapy was used to treat this condition.

ELIGIBILITY:
Inclusion Criteria:

* FA revealed many aneurysms with leakage in the temporal mid-peripheral retina and near the macula. Optical coherence tomography (OCT) showed moderate to marked cystoid macular edema and subretinal fluid. There were no abnormal findings in the cornea, anterior chamber, or lens. No particular lesions were found in the opposite eye of each subject. Based on these findings, the patients were diagnosed with Leber's miliary aneurysm.

Exclusion Criteria:

-

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2021-03-29 (Estimated); Study Completion 2021-05-29 (Estimated)

PRIMARY OUTCOMES:
Visual acuity improvement | 6 months after 3 consequative injections

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided